CLINICAL TRIAL: NCT01478945
Title: Pilot Randomised Controlled Trial of Hand Held NB-UVB for the Treatment of Focal or Early Vitiligo at Home
Brief Title: HI-Light Pilot Trial for Vitiligo: Hand Held NB-UVB for Early or Focal Vitiligo at Home
Acronym: HI-Light
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 11/EM/0331; PR-PG-040710177 (Other Grant/Funding Number: NIHR "SPRUSD" grant)
Record Dates: First submitted 2011-11-15; First posted 2011-11-23 (Estimated); Last update posted 2013-08-23 (Estimated); Status verified 2013-08

CONDITIONS: Vitiligo
Keywords: vitiligo; early vitiligo; focal vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dermfix 1000 active 311 nm NB-UVB (Active Comparator): Active hand held NB-UVB unit:
  Manual device administering NB-UVB
  Interventions: Device: 311 nm NB-UVB light
- Waldmann active 311 nm NB-UVB (Active Comparator): Active hand held NB-UVB unit:
  Manual device administering NB-UVB (Waldmann)
  Interventions: Device: 311 nm NB-UVB light
- Dermfix 1000 placebo (Sham Comparator): Manual placebo hand held NB-UVB unit
  Interventions: Device: 311 nm NB-UVB light

INTERVENTIONS:
Device: 311 nm NB-UVB light — Narrowband UVB is now the most common form of phototherapy used to treat skin diseases. Narrow-band refers to a specific wavelength of ultraviolet (UV) radiation, 311 to 312 nm. Hospital NB-UVB usually involves whole body cabinets suitable for extensive, generalised vitiligo i.e. large or multiple lesions. Usually the whole body is exposed to the UVB for a short time (seconds to minutes). NB-UVB is also used in the treatment of many other skin conditions including psoriasis and eczema.
  Hand held phototherapy units use the same lamp as the whole body units (TLO1) but only suitable for the treatment of smaller areas of skin i.e. early and focal lesions of vitiligo.
  Early reports showed that these units are also safe and effective for the treatment of psoriasis of the scalp.
  Other Names: NB-UVB UV NB 311 UVTLO1

SUMMARY:
This study is a small pilot randomised controlled trial (RCT) comparing hand-held NB-UVB light devices with placebo devices. These devices will be used by the participants to treat their vitiligo at home for a period of four months. The main purpose of the trial is to provide feasibility data that can be used to inform the design of a future multi-centre RCT of these devices. Two hand-held UVB devices with similar manual operating system are being tested during this pilot study. This trial will help the investigators to establish which device is likely to be best for the main trial.

Participants will be approached in a variety of ways (through secondary care, primary care and through direct advertising). Potential participants who contact the co-ordinating centre expressing an interest in the trial will be given more information about the trial, checked for preliminary eligibility, and sent an appointment for a screening visit at the closest recruiting hospital (Nottingham or Leicester).

This screening visit will be conducted by a research nurse, but a dermatologist will also be present in order to confirm the diagnosis of vitiligo and to confirm the participant's suitability for UVB treatment at home. If eligible and willing to take part in the trial, participants will provide written informed consent and baseline data will be collected. In order to define the starting dose to be used when treating the vitiligo, a minimum erythema dose (MED) test will be conducted.

An educational session will be provided by the research nurse outlining how to use the devices, how to assess side-effects of the treatment and how to complete the treatment diary. It is anticipated that the screening visit and educational session will take place on the same day and may take up to 1.5 hours.

On the following day, a brief visit to the hospital will be required in order to examine the skin and read the MED results (if more convenient, the educational session may be delivered at this time). Once this has been done, participants will be given the devices to use at home - treatment is applied 3 times per week on alternate days. They will be followed up by telephone at week 1, week 2 and week 12 - in order to provide support and to monitor side-effects. Participants will be asked to keep a treatment diary that records when the treatment has been used and records side-effects experienced. Emergency contact details will be provided in case of urgent medical need.

Participants will continue with treatment at home for the 16-week trial period. Two further hospital visits will take place in order to record outcome data

DETAILED DESCRIPTION:
This study is a pilot trial to determine the feasibility of conducting a subsequent large multi-centre RCT.

The objectives of this pilot trial are:

Primarily:

1. To establish the proportion of eligible participants and their willingness to be randomised to home NB-UVB

   Secondarily:
2. To establish participants' adherence and satisfaction in using home phototherapy
3. To assess success of blinding of both participants and outcome assessors by using an identical placebo unit with visible light fluorescence bulb instead of NB-UVB bulb.
4. To establish possible short term side effects i.e. if the device is suitable for home use with limited medical supervision
5. To manualise the treatment intervention, i.e. prepare package educating participants in how to use the intervention and to deal with possible side effects.
6. To define and test the primary and secondary outcome measures and the methods of data collection for the main RCT

Trial Configuration:

Parallel groups-Three arms study

1. Group A: active hand held NB-UVB unit (Dermfix 1000)
2. Group B: active hand held NB-UVB unit (Waldmann)
3. Group C: placebo hand held NB-UVB unit (placebo Dermfix 1000) The allocation to the active or placebo group will be 2:1. This trial configuration will reflect the participants' allocation to active and placebo groups in the main RCT (75% of the participants will receive active treatment), as the latter is most likely to be a three arm or a factorial trial. Subsequently, the results obtained from this pilot trial regarding the participants' willingness to be randomised will be a more precise estimate of the main RCT.

Setting:

Participants will primarily be indentified in secondary care (Nottingham, Leicester, Derby and Mansfield) and by direct advertising. Recruitment will be extended to include primary care if time and resources allow.

Sample size estimate:

This is a pilot study, with sample size being resource driven in terms of available subjects in a reasonable time frame, for which no formal statistically based sample size estimate is applicable.

For this pilot study, 21 participants (7 in each group) will allow the investigators to measure the recruitment rate from each site; n=21 will also give a reasonable estimate of acceptability and completeness of outcome data.

Number of participants:

The investigators estimate to recruit 21 participants, 7 in each group; however the recruitment will depend on time and resources available.

Description of interventions:

The hand held NB-UVB unit is a portable and light weight NB-UVB device that is slightly larger than a usual hairbrush.

These units are CE marked and are being used within their licensing authorisations.

The hand held device is held above any small area of the skin (10-12cm x 6.5-4 cm) and spacers are provided in order to standardise the distance from the skin. Hand held NB-UVB units are suitable for small lesions making phototherapy available for participants with limited disease, and for participants who find it difficult to attend hospital-based phototherapy units 2 to 3 times a week.

The lamp is held still above the vitiliginous lesion. If the size of the lesion is bigger than mentioned above i.e. 10-12 cm X 6.5-4 cm, the participant (or their parent or legal guardian for younger participants) will be asked to move the lamp slowly above the area in circular movements.

In this trial the investigators will explore 2 similar hand held NB-UVB (311nm) phototherapy devices with the same output, but a slighly different size of treatment window, weight of the device and cable length. By doing this the investigators will be able to monitor and assess which of the 2 units is best tolerated in terms of participants' satisfaction and minimisation of side effects. The information gathered will assist in the choice of device for the main RCT.

Device A: Dermfix 1000 NB-UVB Device B: Waldmann UV 109 Both devices are manual units with an on/off switch and an external digital timer. The user of this device has to follow the written treatment protocol, set and re-set the timer each time manually and to keep an accurate diary of exposure times.

The devices need to be connected to a socket all the time.

Placebo Device: Placebo Dermfix 1000, same as Device A The placebo device to be used is identical to the active device Dermfix with the only difference that it will not emit 311nm NB-UVB.

Duration of study:

The recruitment is planned to commence as soon as approvals (ethics and R&D) are in place and should take approximately 6 months. Each participant will participate in the study for 4 months. Participants will be assessed at face to face visits at the beginning of the screening stage-baseline, 8th week and 16th week. Outcomes will be assessed at the same time points.

Follow up telephone calls will be made at weeks 1, 2 and 12.

Randomisation and blinding:

Participants will be blinded to which device they have received, (intervention groups A or B or control group C).

The research nurse will be blinded to which group the participants are allocated (intervention groupS A or B or control group C).

The randomisation will be based on a computer generated pseudo-random code using random permuted blocks of randomly varying size, created by the Nottingham Clinical Trials Unit (CTU) in accordance with their standard operating procedure (SOP) and held on a secure server. The randomisation will be stratified by 3 groups (Group A, B and C) and 2 recruiting sites.

Statistical methods:

Demographic, baseline data and measure of compliance will be summarised by descriptive statistics (number[n], mean, standard deviation [SD], median, minimum and maximum) or frequency tables, stratified by treatment.

Also, calculation of the re-pigmentation rate, spread & cessation of the vitiligo lesions will be conducted for all of the 3 devices. This information will be vital for the sample size calculation for the definitive trial.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a diagnosis of vitiligo confirmed by dermatologist. Participants with focal disease, less than 25% of body surface area.
* Age: children and adults (no upper age limit). The child has to be older than 5 years old and/or mature enough to understand that the eyes must be kept closed, and to stay still for the duration of treatment.
* No therapy for vitiligo in the previous 2 weeks and no other vitiligo treatment during the trial other than as per trial protocol.
* Participants with both spreading and stable disease
* Participants able to give informed consent. We will aim to treat all vitiligo lesions, however the participant (and parent/legal guardian if the participant is a child) and research nurse will agree at the beginning of the trial if there are any lesions participants would not want to be treated, such as on non exposed sites or areas difficult to reach to treat, e.g. back.

Exclusion Criteria:

* Segmental vitiligo
* Universal vitiligo
* Previous history of skin cancer
* Recent or concurrent radiotherapy
* Photosensitivity
* Use of immunosuppressive or photosensitive drugs
* Pregnant or lactating women
* Any major medical co-morbidities
* Vitiligo lesions on genitalia should not be treated

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2012-02; Primary Completion 2012-09 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Proportion of eligible participants, willing to be randomised. | 4 to 6 months
  To establish the proportion of eligible participants and their willingness to be randomised to home NB-UVB

SECONDARY OUTCOMES:
Number of participants accepting the initial invitation to participate | 4 to 6 months
Proportion of participants fulfilling trial eligibility criteria | 4 to 6 months
Proportion of participants adhering to the treatment protocol | 4 months
  To establish participants' adherence in using home phototherapy
Proportion of participants (or their parent/legal guardian) who are satisfied with the treatment and the hand held units. | 4 months
  To establish participants' satisfaction in using home phototherapy
Proportion of participants for whom the blinding of the assessor and the allocated group is maintained | 4 months
  To assess success of blinding of both participants and outcome assessors by using an identical placebo unit with visible light fluorescence bulb instead of NB-UVB bulb.
Incidence of NB-UVB short term adverse events | 4 months
  To manualise the treatment intervention, i.e. prepare package educating participants in how to use the intervention and to deal with possible side effects.
  To establish possible short term side effects i.e. if the device is suitable for home use with limited medical supervision
Outcome measures for the main large trial will also be tested. These will include: repigmentation rate of vitiliginous lesions, cessation of spreading of vitiligo, impact on the quality of life of participants. | 4 months
  To define and test the primary and secondary outcome measures and the methods of data collection for the main RCT

CONTACTS AND LOCATIONS:
Overall Officials: Hywel C. Williams, MSc PhD FRCP, Study Chair — Centre of Evidence Based Dermatology; Viktoria Eleftheriadou, MD, Study Director — Centre of Evidence Based Dermatology; Jane C Ravenscroft, MB ChB, MRCP, Principal Investigator — Queen's Medical Center; Anton Alexandroff, PhD MRCP, Principal Investigator — University Hospitals, Leicester
Locations (2):
- United Kingdom (2):
  - Queens Medical Centre,Nottingham University Hospitals NHS Trust, Nottingham, East Midlands
  - Leicester Royal Infirmary, Leicester, Leicestershire

REFERENCES:
- [Background] Whitton ME, Pinart M, Batchelor J, Lushey C, Leonardi-Bee J, Gonzalez U. Interventions for vitiligo. Cochrane Database Syst Rev. 2010 Jan 20;(1):CD003263. doi: 10.1002/14651858.CD003263.pub4. PMID 20091542
- [Background] Gonzalez U, Whitton M, Eleftheriadou V, Pinart M, Batchelor J, Leonardi-Bee J. Guidelines for designing and reporting clinical trials in vitiligo. Arch Dermatol. 2011 Dec;147(12):1428-36. doi: 10.1001/archdermatol.2011.235. Epub 2011 Aug 15. PMID 21844427
- [Background] Gawkrodger DJ, Ormerod AD, Shaw L, Mauri-Sole I, Whitton ME, Watts MJ, Anstey AV, Ingham J, Young K. Vitiligo: concise evidence based guidelines on diagnosis and management. Postgrad Med J. 2010 Aug;86(1018):466-71. doi: 10.1136/pgmj.2009.093278. PMID 20709768
- [Background] Eleftheriadou V, Whitton ME, Gawkrodger DJ, Batchelor J, Corne J, Lamb B, Ersser S, Ravenscroft J, Thomas KS; vitiligo priority setting partnership. Future research into the treatment of vitiligo: where should our priorities lie? Results of the vitiligo priority setting partnership. Br J Dermatol. 2011 Mar;164(3):530-6. doi: 10.1111/j.1365-2133.2010.10160.x. Epub 2011 Jan 28. PMID 21128908
- [Derived] Eleftheriadou V, Thomas K, Ravenscroft J, Whitton M, Batchelor J, Williams H. Feasibility, double-blind, randomised, placebo-controlled, multi-centre trial of hand-held NB-UVB phototherapy for the treatment of vitiligo at home (HI-Light trial: Home Intervention of Light therapy). Trials. 2014 Feb 8;15:51. doi: 10.1186/1745-6215-15-51. PMID 24507484